CLINICAL TRIAL: NCT06615557
Title: US, Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of Fasedienol Nasal Spray for the Acute Treatment of Anxiety Induced by a Public Speaking Challenge in Adult Subjects With Social Anxiety Disorder, With an Open-Label Extension (PALISADE-4)
Brief Title: Fasedienol Nasal Spray for the Acute Treatment of Anxiety in Adults With Social Anxiety Disorder (PALISADE-4)
Acronym: PALISADE-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH94B-CL043
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Social Anxiety Disorder (SAD)
Keywords: Fasedienol; PH94B; social anxiety disorder; social anxiety; SAD; pherine; pherine nasal spray; acute treatment; anxiolytic; mental health; anxiety; performance anxiety; anxiety nasal spray; anxiety treatment; public speaking anxiety; social phobia; phobic disorders; mental disorder; speech task
MeSH Terms: conditions — Phobia, Social; Psychological Well-Being; Anxiety Disorders; Phobic Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasedienol Nasal Spray (Experimental)
  Interventions: Drug: Fasedienol Nasal Spray
- Placebo Nasal Spray (Experimental)
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: Fasedienol Nasal Spray — Nasal spray delivered 20 minutes before the PSC
  Arms: Fasedienol Nasal Spray
Drug: Placebo Nasal Spray — Nasal spray delivered 20 minutes before the PSC
  Arms: Placebo Nasal Spray

SUMMARY:
This U.S. Phase 3 clinical trial is designed to evaluate the efficacy, safety, and tolerability of the acute intranasal (i.n.) administration of Fasedienol Nasal Spray (fasedienol) (3.2 µg) to relieve symptoms of acute anxiety in adult subjects ages 18 through 65 with Social Anxiety Disorder induced by a public speaking challenge (PSC) in a clinical setting. In addition, safety and tolerability of i.n. administration of 3.2 µg of fasedienol, as-needed, up to 6 times per day for up to 12 months, will be assessed in those subjects who complete PALISADE-4 and choose to enter the distinct open-label extension phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided prior to conducting any study-specific assessment.
* Male and female adults, 18 through 65 years of age, inclusive.
* Current diagnosis of SAD as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, and confirmed by the Mini-International Neuropsychiatric Interview (MINI).
* Clinician-rated Liebowitz Social Anxiety Score (LSAS) total score ≥70 at Screening (Visit 1).
* Clinician-rated Hamilton Depression Rating Scale (HAM-D) (17-items) total score <16.
* Female subjects of childbearing potential must be able to commit to the consistent and correct use of an effective method of birth control throughout the study
* Subjects must have normal olfactory function

Exclusion Criteria:

* Any history of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, psychosis, anorexia or bulimia, premenstrual dysphoric disorder, autism spectrum disorder, or obsessive-compulsive disorder.
* Any other current principal or personality disorder (previously known as Axis I or Axis II disorders), except for specific phobias or generalized anxiety disorder, provided that these are not the primary diagnosis.
* Subjects who meet criteria for moderate or severe alcohol use disorder within the 1 year prior to study entry, or any use of illicit substances or tetrahydrocannabinol ("THC") within 2 months prior to study entry.
* In the opinion of the investigator, the subject has a significant risk for suicidal behavior during the course of their participation in the study, or the subject is considered to be an imminent danger to themself or others.
* Clinically significant nasal pathology or history of significant nasal trauma, nasal surgery, total anosmia, or nasal septum perforation that may have damaged the nasal chemosensory epithelium.
* Two or more documented failed adequate treatment trials with a registered medication approved for SAD.
* Currently receiving cognitive-behavioral therapy (CBT), exposure therapy, or acceptance and commitment therapy.
* Subjects taking psychotropic medications within 30 days before Visit 2.
* Use of any over-the-counter product, prescription product, off-label treatment, cannabidiol ("CBD"), or herbal preparation for treatment of the symptoms of anxiety or social anxiety within 30 days before Visit 2.
* Prior participation in a clinical trial involving fasedienol.
* Participation in any other clinical trial within the last 30 days or during the course of the current trial.
* Subjects with a positive urine drug screen.
* Women who have a positive urine pregnancy test.
* Women who are currently breastfeeding are not eligible unless they are willing to stop breastfeeding for the duration of the study.
* Subjects who have tested positive and/or have exhibited symptoms consistent with SARS-CoV-2 infection during the 4 weeks prior to Screening (Visit 1).
* Any clinically significant medical history or findings as determined by the Investigator that could interfere with the objectives of the study or put the participant at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | 7 days (Visit 2 to Visit 3)
  The SUDS is a patient self-rated scale that is scored in the range of 0 to 100 (operationalized for participants in this study as 0=totally relaxed or no anxiety and 100=highest distress or anxiety ever felt).

SECONDARY OUTCOMES:
Global Impression Scale of Improvement (CGI-I) | 7 days (Visit 2 to Visit 3)
  The CGI-I scale is a clinician-rated scale to assess illness improvement. The CGI-I scale includes one item being scored from 1 (best outcome) to 7 (worst outcome) with 4 being no change.
Patient Global Impression of Change (PGI-C) | 7 days (Visit 2 to Visit 3)
  The PGI-C is a patient self-rated scale to assess improvement. The PGI-C includes 7 items being scored from 1 (best outcome) to 7 (worst outcome) with 4 being no change.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Vistagen Clinical Site, Phoenix, Arizona
  - Vistagen Clinical Site, Little Rock, Arkansas
  - Vistagen Clinical Site, Bellflower, California
  - Vistagen Clinical Site, Oceanside, California
  - Vistagen Clinical Site, Orange, California
  - Vistagen Clinical Site, Redlands, California
  - Vistagen Clinical Site, Torrance, California
  - Vistagen Clinical Site, Denver, Colorado
  - Vistagen Clinical Site, Tampa, Florida
  - Vistagen Clinical Site, Decatur, Georgia
  - Vistagen Clinical Site, Chicago, Illinois
  - Vistagen Clinical Site, Naperville, Illinois
  - Vistagen Clinical Site, Boston, Massachusetts
  - Vistagen Clinical Site, Bloomfield Township, Michigan
  - Vistagen Clinical Site, Flowood, Mississippi
  - Vistagen Clinical Site, Las Vegas, Nevada
  - Vistagen Clinical Site, Albuquerque, New Mexico
  - Vistagen Clinical Site, New York, New York
  - Vistagen Clinical Site, Cincinnati, Ohio
  - Vistagen Clinical Site, Austin, Texas
  - Vistagen Clinical Site, Dallas, Texas
  - Vistagen Clinical Site, Houston, Texas
  - Vistagen Clinical Site, San Antonio, Texas
  - Vistagen Clinical Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://socialanxietytrials.com/